CLINICAL TRIAL: NCT02758548
Title: A Multicenter Clinical Evaluation Study to Determine the External Site Accuracy of Total Immunoglobulin E Measurement Using a Novel Point of Care Test Device Compared to a Reference Method in Atopic Subjects
Brief Title: Determination of Accuracy in Measurement of Total Immunoglobulin E Using a Test Device in Atopic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDIGE0012201
Record Dates: First submitted 2016-03-15; First posted 2016-05-02 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Atopic Asthma
Keywords: Total IgE measurement; Novel Point-of-care test device; atopic conditions; in vitro diagnostic test
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capillary Blood Sampling (Other): Capillary blood sampling, collected as two fingerprick samples with POCT device and two venous samples
  Interventions: Procedure: Blood sample; Device: POCT device

INTERVENTIONS:
Procedure: Blood sample — Fingerprick and venous
Device: POCT device — Investigational device

SUMMARY:
The purpose of this study is to determine the accuracy of the Novel point of care test (POCT) total IgE assay in atopic patients.

120 patients with atopic conditions and approximately 40 healthy subjects will be enrolled. Fingerstick capillary blood samples will be collected and tested in the POCT device. Venous samples will be collected and sent to a reference laboratory for measurement of serum total IgE using the reference immunoassay method.

ELIGIBILITY:
Inclusion criteria: atopic patients

* Subjects who are diagnosed with atopic condition
* Subjects or legal guardians who are able to give informed consent
* Other protocol-defined inclusion criteria may apply Exclusion criteria: atopic patients
* Subjects who have received anti-IgE antibody treatment
* Subjects who have elevated IgE levels for reasons other than allergic conditions
* Other protocol-defined exclusion criteria may apply Inclusion criteria: healthy subjects
* Subjects who are able to give informed consent for participation in the study according to local requirements / law.

Exclusion criteria: healthy subjects

* Subjects who have received anti-IgE antibody treatment
* Subjects with a suspected or confirmed clinical diagnosis of an atopic condition
* Other protocol-defined exclusion criteria may apply

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Total IgE concentration | Day 0 or Day 1 (Visit 2: Blood sampling)
  Total IgE concentration in capillary blood measured with the POCT device at Day 0 or Day 1 from enrollment.
  Total IgE concentration in venous blood measured with the reference method at Day 0 or Day 1 from enrollment.

SECONDARY OUTCOMES:
Device usability questionnaire response | Day 0 or Day 1 (Visit 2: Blood sampling)
  Device usability assessment of the POCT device as per operators at the completion of the study.

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (2):
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Lübeck
- Italy (3):
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
- Netherlands (2):
  - Novartis Investigative Site, Harderwijk, Netherlands
  - Novartis Investigative Site, Almelo
- Spain (2):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Valencia, Valencia
- United Kingdom (3):
  - Novartis Investigative Site, Chertsey, Surrey
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Manchester